CLINICAL TRIAL: NCT04472663
Title: Patient Reported Outcomes And Treatment Experiences In Renal Cell Carcinoma (ONE-RCC)
Brief Title: Participant Reported Outcomes and Treatment Experiences in Kidney Cancer
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-7DK
Record Dates: First submitted 2020-07-14; First posted 2020-07-15 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-01

CONDITIONS: Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1: Retrospective Long-term Chart Review
- Cohort 2: Prospective-Retrospective Chart Review and Humanistic Burden

SUMMARY:
The purpose of this observational study is to collect contemporary real-world treatment patterns, clinical outcomes, humanistic burden (including patient-reported disease-specific Health-related Quality of Life (HRQoL), and treatment- related adverse events (AEs) or adverse reactions (ARs) among Advanced Renal Cell Carcinoma (aRCC) patients initiating first-line systemic therapy.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

Cohort 1

* Primary diagnosis of aRCC (advanced Renal Cell Carcinoma) or metastatic RCC
* Medical history must be available from date of aRCC diagnosis
* Initiated 1LOT between April 2018 - March 2020

Cohort 2:

* Primary diagnosis of aRCC (not amenable to curative surgery or radiation therapy/ AJCC Stage III unresectable) or metastatic RCC (AJCC Stage IV).
* Medical history must be available from date of aRCC diagnosis.
* Initiate 1LOT.

Exclusion Criteria:

* Currently enrolled in a clinical trial for treatment of aRCC
* Any prior malignancy active within the previous 3 year, except for locally curable cancers that have been cured
* Any prior systemic therapy for aRCC, with the exception of neoadjuvant or adjuvant therapy (Cohort 2 only)

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be included if they have primary diagnosis of aRCC, age ≥18 years, with medical history available from date of aRCC diagnosis to most recent or current therapy. For Cohort 1, patients will be eligible if they had initiated 1LOT between April 2018 - March 2020. For Cohort 2, patients will be eligible if they are about to initiate 1LOT, must be willing to sign the informed consent form (ICF), where required, and complete the humanistic burden assessment at baseline and subsequent follow-ups.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2020-12-09 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 36 months
Disease-related symptoms as measured by change from baseline in FKSI-DRS | Up to 36 months

SECONDARY OUTCOMES:
Demographic characteristics of aRCC patients as measured by continuous statistics: Age | Up to 36 months
Demographic characteristics of aRCC patients as measured by categorical statistics: Gender | Up to 36 months
Demographic characteristics of aRCC patients as measured by categorical statistics: Race/ethnicity | Up to 36 months
Demographic characteristics of aRCC patients as measured by continuous statistics: Height | Up to 36 months
Demographic characteristics of aRCC patients as measured by continuous statistics: Smoking status | Up to 36 months
Demographic characteristics of aRCC patients as measured by continuous statistics: Family history of RCC | Up to 36 months
Demographic characteristics of aRCC patients as measured by continuous statistics: Healthcare coverage (medical and drug) | Up to 36 months
Sequence of therapy events including treatment modalities | Up to 36 months
Time to therapy initiation of LOT | Up to 36 months
Rationale for therapy selection | Up to 36 months
Switching and/or discontinuation rate | Up to 36 months
Drug use characteristics including dosing regimens: Drugs included in each course of therapy | Up to 36 months
Drug use characteristics including dosing regimens : Formulations | Up to 36 months
Drug use characteristics including dosing regimens : Dose | Up to 36 months
Drug use characteristics including dosing regimens : Frequency of administration | Up to 36 months
Drug use characteristics including dosing regimens: Duration of therapy | Up to 36 months
Drug use characteristics including dosing regimens : Number of cycles planned and administered | Up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Morristown, New Jersey, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm